CLINICAL TRIAL: NCT03967275
Title: Subconjunctival Injection of Allogeneic Mesenchymal Stem Cells in Severe Ocular Chemical Burn SyMbOL Pre Clinical Study
Brief Title: Subconjunctival Injection of Allogeneic Mesenchymal Stem Cells in Severe Ocular Chemical Burn
Acronym: SYMBOLpreclini
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: EGN_2018_11
Record Dates: First submitted 2019-05-26; First posted 2019-05-30 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Bone Marrow Donor
Keywords: Bone marrow harvest; Bone Marrow derived Mesenchymal Stem Cells (BM-MSC); Pre-clinical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: bone marrow harvest — During bone marrow harvest, an additional 10 mL sample will be collected for the study.

SUMMARY:
The objective of this pre-clinical study is to demonstrate the robustness of Bone Marrow derived Mesenchymal Stem Cells (BM-MSC) production, to treat patients with severe eye burns.

For bone marrow donors who agree to participate, a 10 ml BM sample will be collected apart the 1 liter BM dedicated to transplantation.

A maximum of three donors of allogeneic BM-MSCs will be included. A ready-to-use BM-MSC suspension will be produced and stored for 10 years to accumulate data about stability of cryopreserved cells.

ELIGIBILITY:
Inclusion criteria:

- Patient with a bone marrow donation planned

Exclusion criteria:

* The donor is finally not eligible
* The harvest cannot be performed
* The sample cannot be obtained during the BM harvest procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bone marrow donors
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
The number of donors needed to obtain 3 BM harvest. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis Hospital, APHP, Paris, France

IPD SHARING:
Plan to Share IPD: No